CLINICAL TRIAL: NCT01533870
Title: An Open-label, Fixed-sequence, 3-period, 3-treatment, Crossover Study to Assess the Effects of Rifampin on Pharmacokinetics of NKTR-118 in Healthy Subjects
Brief Title: Study in Healthy Volunteers to Investigate the Effects of Rifampin on the Pharmacokinetics of NKTR-118
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D3820C00015
Record Dates: First submitted 2012-02-13; First posted 2012-02-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Drug Induced Constipation
Keywords: Phase 1; Healthy male and female volunteers; Drug-drug interaction; Pharmacokinetics; NKTR-118; Bioavailability; Plasma AUC and Cmax; Plasma AUC0-t and t1/2λz and tmax
MeSH Terms: interventions — naloxegol; Rifampin

ARMS (3):
- NKTR-118 (Experimental): Single dose NKTR-118 25 mg on Day 1 only
  Interventions: Drug: NKTR-118
- Rifampin (Active Comparator): Rifampin 600 mg once daily on Days 4 to 12
  Interventions: Drug: Rifampin
- Rifampin/ NKTR-118 (Active Comparator): Rifampin 600 mg plus NKTR-118 25 mg on Day 13
  Interventions: Drug: NKTR-118; Drug: Rifampin

INTERVENTIONS:
Drug: NKTR-118 — Oral 25 mg
  Arms: NKTR-118; Rifampin/ NKTR-118
Drug: Rifampin — Oral 600 mg
  Arms: Rifampin; Rifampin/ NKTR-118

SUMMARY:
Study in healthy volunteers to investigate the effects of Rifampin on the Pharmacokinetics of NKTR-118.

DETAILED DESCRIPTION:
An Open-label, fixed-sequence, 3-period, 3-treatment, Crossover Study to Assess the Effects of Rifampin on Pharmacokinetics of NKTR-118 in Healthy Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study-specific procedures.
* Male and female (nonchildbearing potential, nonlactating) healthy volunteers aged 18 to 55 years inclusive, with suitable veins for cannulation or repeated venipuncture.
* Female volunteers must have a negative pregnancy test at screening and at admission, must not be lactating, and must be of nonchildbearing potential.
* Male volunteers should be willing to use barrier contraception ie, condoms, from the first day of dosing until 3 months after dosing with the IP. The female partner should use contraception during this period.
* Volunteers must have a BMI between 18 and 30 kg/m2, inclusive, and weigh at least 50 kg.

Exclusion Criteria:

* Any clinically significant disease or disorder (eg, cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, or major physical impairment), as judged by the Investigator.
* Any clinically significant illness, medical/surgical procedure or trauma, in the opinion of the Investigator, within 4 weeks of the first administration of IP.
* Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results as judged by the Investigator.
* Significant orthostatic reaction at enrollment as judged by the Investigator.
* Abnormal vital signs, after 10 minutes supine rest as defined in protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Description of the pharmacokinetic(PK) profile for NKTR 118 after co administration of Rifampin in terms of area under the concentration-time curve from time zero (predose) extrapolated to infinity (AUC). | Predose and at 0:15, 0:30, 1, 1:30, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours Day 1 and 13
Description of the PK profile for NKTR 118 in terms of maximum plasma concentration (Cmax), time to Cmax (tmax), half-life (t1/2λz), apparent terminal rate constant (λz). | Predose and at 0:15, 0:30, 1, 1:30, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours Day 1 and 13
Description of the PK profile for NKTR 118 in terms of area under the plasma concentration-time curve from time zero to the time of the last measurable concentration [AUC(0-t)]. | Predose and at 0:15, 0:30, 1, 1:30, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours Day 1 and 13
Description of the PK profile for NKTR 118 in terms of area under the plasma concentration-time curve from time zero to 24 hours [AUC(0-24)]. | Predose and at 0:15, 0:30, 1, 1:30, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours Day 1 and 13
Description of the PK profile for NKTR 118 in terms of apparent oral clearance (CL/F), and apparent volume of distribution during the terminal phase (Vz/F). | Predose and at 0:15, 0:30, 1, 1:30, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours Day 1 and 13

SECONDARY OUTCOMES:
Description of the safety profile in terms of adverse events, clinical laboratory assessments , vital signs (blood pressure and pulse rate), physical examinations, electrocardiograms, and Columbia-Suicide Severity Rating scale. | From baseline day -1 through to Follow-up (Maximum 27 days)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Fransson, MD, Study Chair — AstraZeneca, Sodertalje Sweden; Kelli Craven, MD, Principal Investigator — Quintiles, Inc Kansas Overland Park US.; Mark Sostek, MD, Study Director — AstraZeneca, Wilmington US
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1396&filename=D3820C00015.pdf